CLINICAL TRIAL: NCT01935466
Title: Pioglitazone and Risk of Bladder Cancer in Patients With Type 2 Diabetes Mellitus"PROBE-PIO"Study
Brief Title: Risk of Bladder Cancer in Type 2 Diabetes Patients With Pioglitazone Therapy "PROBE"
Acronym: PROBE-PIO
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ashu Rastogi, Assisstant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: PROBEPIO
Record Dates: First submitted 2013-08-22; First posted 2013-09-05 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Bladder Cancer
Keywords: Pioglitazone; Bladder cancer; Type 2 Diabetes
MeSH Terms: conditions — Urinary Bladder Neoplasms; Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pioglitazone: Ever users of Pioglitazone
  Interventions: Drug: Pioglitazone
- Other drugs: Never users of pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Ever users of Pioglitazone
  Other Names: Pioglit,; Pioz
  Groups: Pioglitazone

SUMMARY:
Pioglitazone, an agonist of the peroxisome-proliferator-activated receptor (PPAR), is a relatively new oral anti-hyperglycemic drug. Since its first approval in the USA in 1999, a potential link with bladder cancer has been a subject of debate. US Food and Drug Administration (FDA) in September, 2010 and European Medicines Agency in July, 2011 issued an alert about a potential relation between the occurrence of bladder cancer and the prescription of pioglitazone, based on the data from various studies. France banned its use in July 2011.

Recently Pioglitazone was banned from India without any evidence of increased bladder cancer in our population. With this background, we plan to study the risk of bladder cancer in male type 2 diabetes subjects aged more than 50 years who are on pioglitazone therapy as compared to never-users of pioglitazone in a retrospective cohort design and provide the first data from India to the policy makers regarding the purported risk in our ethnicity and geographical area.

DETAILED DESCRIPTION:
Very recently, pioglitazone was banned for use in type 2 diabetes patients in India as well, by the notification from Government of India based on a case series - the ban was revoked a few days later due to lack of evidence.

The incidence rates of bladder cancer among different ethnicities differ markedly, with Caucasians having the highest incidence. Another important distinction pertains to the dose of pioglitazone- the daily dose of pioglitazone used in the previous studies (from western countries) was 45 mg, which is higher than currently prescribed in India (7.5-30 mg). Therefore the risk of bladder cancer in Indian patients cannot be extrapolated from studies conducted in other regions of the world. Consequently, it is an interesting issue to explore the risk of bladder cancer amongst the pioglitazone-users in our settings with different ethnicity and risk profile. There has been a single report of eight cases of sporadic bladder cancer from India.10 However, the study had no denominator and there has been no further study from India exploring the relationship between pioglitazone and bladder cancer.

Furthermore the risk of bladder cancer is highest in males greater than 50 years. The other risk factors are smoking, occupational exposure to aromatic amines in metal, leather, and paint industries etc., all of which are more common in males. The increase, if any, in the rate of bladder cancer with pioglitazone is expected to be highest in this group.

The results from currently available studies either in-vitro, animal, human (observational) on the link between pioglitazone and bladder cancer are not consistent. Whether the positive link in patients using pioglitazone in some studies could be due to the drug per se, or due to the underlying disease of diabetes, the interactions with other concomitant drugs, the inherent flaws associated with study designs and statistical analyses, or the different ethnicities between studies, are worthy of discussion. Diabetes per se may increase the risk of cancer, probably via the activation of the Ras/Raf mitogen-activated protein kinase pathway in association with a reduction of the expression of epidermal growth factor receptor. In fact, epidemiologic studies also suggest an increased risk of bladder cancer in diabetic patients, independent of the commonly used oral anti-diabetic agents or insulin.

Hence we plan to investigate the risk of bladder cancer in type 2 diabetes subjects using pioglitazone as compared to those who have never been exposed to pioglitazone. We will thoroughly scrutinize the records and also interview the subjects regarding other risk factors for bladder cancer in addition to pioglitazone.

ELIGIBILITY:
Inclusion Criteria:

1. Male Type 2 diabetes subjects with age >50 year
2. On anti-diabetic drugs and/or insulin for≥ 1 year
3. Patient willing to provide informed consent to be included in the study

Exclusion Criteria:

* 1. Bladder cancer diagnosed before the onset of Diabetes mellitus. 2. Patient not willing to participate in the study.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group will comprise of male type 2 diabetes subjects having used pioglitazone for one year or more. The control group will include male type 2 diabetes subjects on medications other than pioglitazone adjusted for age, household income, anti-diabetic drugs, HbA1c,smoking, renal function and other bladder disorders.
Sampling Method: Non-Probability Sample
Enrollment: 6107 (Actual)
Dates: Start 2013-07; Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Bladder cancer rate | Prevalent bladder cancer on pioglitazone or anti diabetic drugs for 1 year
  Kaplan-Meir survival curves will be generated for the two groups of pioglitazone users and non-pioglitazone users. All the data at the time point of interview will be considered censored. Bladder cancer rates among pioglitazone users and non-users will be compared by hazard ratio (HR) after Cox regression. Adjustment for various confounders like age, diabetes duration, region of residence, occupation, smoking, urinary tract disease, use of other medications like sulfonylurea, metformin, insulin, DPP-IV inhibitors and other cancers before baseline would be done.

CONTACTS AND LOCATIONS:
Locations (1):
- Deptt of Endocrinology, Chandigarh, India